CLINICAL TRIAL: NCT06669351
Title: A Multicenter, Randomized, Double-blind, Positive Controlled Phase Ⅲ Clinical Trial of ZX-7101A Tablets to Evaluate the Safety and Efficacy in the Treatment of Uncomplicated Influenza in Children Aged 5-11 Years
Brief Title: Study to Assess the Safety and Efficacy of ZX-7101A in Children Aged 5-11 Years With Influenza
Acronym: ZX-7101A-210
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the company's development strategy.
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX-7101A-210
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Viral Infection
Keywords: influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Part 1:
  A pilot study of pharmacokinetics, safety, and efficacy was conducted in children (5-11 years old, weight ≥20kg) with uncomplicated influenza.
  A total of 12 subjects were planned to be enrolled. (Pharmacokinetic and safety data from at least 8 children are required.)
  Part 2:
  A randomized phase III study with safety as primary endpoint was conducted in children (5-11 years old, body weight ≥20kg) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A or oseltamivir phosphate.
  Enrolled subjects were required to have typical systemic and/or respiratory influenza symptoms, with first influenza symptoms occurring within 48 hours of randomization. A total of 168 subjects were planned to be enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Arm (Experimental): Part 1:
  A pilot study of pharmacokinetics, safety, and efficacy was conducted in children (5-11 years old, weight ≥20kg) with uncomplicated influenza. A total of 12 subjects were planned to be enrolled.
  Interventions: Drug: ZX-7101A
- Oseltamivir phosphate dry suspension: (Active Comparator): Part 2:
  A randomized phase III study with safety as primary endpoint was conducted in children (5-11 years old, body weight ≥20kg) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A (2 tablets，specification：10mg, single dose) or oseltamivir phosphate dry suspension（specification：0.36g）.
  Interventions: Other: Placebo for ZX-7101A tablet; Drug: Oseltamivir phosphate dry suspension
- ZX-7101A (Experimental): Part 2:
  A randomized phase III study with safety as primary endpoint was conducted in children (5-11 years old, body weight ≥20kg) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A (2 tablets，specification：10mg, single dose) or oseltamivir phosphate dry suspension（specification：0.36g）.
  Interventions: Drug: ZX-7101A; Other: Placebo for Oseltamivir phosphate dry suspension:

INTERVENTIONS:
Drug: ZX-7101A — On day1: Take two tablets of ZX-7101A orally once (specification: 10mg/ tablet) with appropriate amount of warm water
  Arms: Single Arm; ZX-7101A
Other: Placebo for ZX-7101A tablet — Placebo for ZX-7101A tablet:
  The appearance and properties of placebo tablets were identical to those of the trial drug ZX-7101A tablets. On Day 1, two placebo for ZX-7101A tablets were taken orally with appropriate warm water.
  Arms: Oseltamivir phosphate dry suspension:
Drug: Oseltamivir phosphate dry suspension — Drug: Oseltamivir phosphate dry suspension:
  From Day1 to Day 5 : Oseltamivir phosphate suspension was orally administered twice a day, dose according to the label.
  Arms: Oseltamivir phosphate dry suspension:
Other: Placebo for Oseltamivir phosphate dry suspension: — Drug: Placebo for Oseltamivir phosphate dry suspension:
  From Day1 to Day 5 : Placebo for Oseltamivir phosphate suspension was orally administered twice a day, dose according to the label.
  Arms: ZX-7101A

SUMMARY:
A multicenter, randomized, double-blind, positive controlled, phase III trial to evaluate the safety and efficacy of ZX-7101A tablets versus oseltamivir phosphate suspension in children aged ≥5 years and < 12 years with uncomplicated influenza.

DETAILED DESCRIPTION:
Part 1:

A pilot study of pharmacokinetics, safety, and efficacy was conducted in children (5-11 years old, weight ≥20kg) with uncomplicated influenza. A total of 12 subjects were planned to be enrolled. (Pharmacokinetic and safety data from at least 8 children are required.) On the first day, ZX-7101A 20 mg tablets, 2 tablets (specification: 10 mg/ tablet) were taken orally. PK samples were collected before and after the first (D1) dose: 1 to 2 h, 4 h, 8 h, 24 h (D2), 96 h (D5), 192 h (D9) and 336 h (D15) after administration.

Part 2:

A randomized phase III study with safety as primary endpoint was conducted in children (5-11 years old, body weight ≥20kg) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A or oseltamivir phosphate.

Enrolled subjects were required to have typical systemic and/or respiratory influenza symptoms, with first influenza symptoms occurring within 48 hours of randomization. The study was divided into a screening/treatment period (D1) and an observation period (approximately 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 1.≥5 to<12 years of age at the time of randomization, males or females.
* 2.Patients in the screening period met the following criteria:

  1. Rapid influenza diagnostic test (RIDT) or polymerase chain reaction (PCR) test positive;
  2. Axillary temperature ≥ 37.5℃ at screening; If taking antipyretics, axillary temperature ≥ 37.5℃ after taking the drug (more than 4 hours).
  3. At least one of influenza -related systemic symptoms is moderate or greater in severity: a. muscle or joint pain, b. fatigue, c. headache, d. fever.
  4. At least one of the influenza-related respiratory symptoms is moderate or greater in severity: a. nasal congestion, b. sore throat, c. cough.
* 3. The first occurrence of influenza symptoms ≤ 48 hours from the time of patient randomization.

  1. Body temperature ≥ 37.5 ℃ (axillary temperature) or 37.5 ℃ (oral temperature) or 38.0 ℃ (rectal or tympanic membrane temperature)for the first time;
  2. Or at least one systemic or respiratory symptom may occur: a. nasal congestion, b. sore throat, c. cough, d. muscle or joint pain, e. fatigue, f. headache, g. fever.
* 4. Both the subject and his/her guardian are volunteer to participate in the study and sign the written informed consent form (ICF), the subject could comply with all the study procedures, complete the subject diary as required (the guardian is allowed to fill in if necessary).

Exclusion Criteria:

* Patients with severe influenza virus infection requiring inpatient treatment. (Meet any one of the following criteria)

  1. Severe cases with one of the following conditions：

     * Persistent high fever for more than 3 days, accompanied by severe cough, purulent sputum, bloody sputum, or chest pain;
     * Fast breathing rate, difficulty breathing, cyanosis of lips;
     * Delayed response, drowsiness, restlessness, and other mental changes or seizures;
     * Severe vomiting, diarrhea, and dehydration symptoms;
     * Concomitant pneumonia;
     * Significant exacerbation of existing underlying diseases;
     * Other clinical situations that require hospitalization.
  2. Critical cases with one of the following conditions (Including but not limited to)：

     * Respiratory failure;
     * Acute necrotizing encephalopathy;
     * Shock;
     * Multiple organ dysfunction;
     * Other serious clinical situations that require monitoring and treatment.
* 2. High risk population for severe cases. (Meet any one of the following criteria):

  1. Accompanied by the following basic diseases and judged by the investigators to be clinically significant, such as lung diseases, liver diseases, kidney diseases, hematological system diseases, heart diseases, neurological and neuromuscular diseases that affect the ability to clear respiratory secretions, metabolic and endocrine system diseases, etc;
  2. Subjects with low immune function, such as malignant tumors, organ or bone marrow transplants, HIV infections, or those who have been taking immunosuppressants for the past 3 months;
  3. Clinical significance of correcting QT interval abnormalities in electrocardiogram display; (QTc>440ms in male or QTc>450ms in female);
  4. Subjects who require long-term use of drugs containing aspirin or salicylates : It is necessary to take medication containing aspirin or salicylate regularly every day for more than 14 days;
  5. BMI exceeds the standards.
* 3. Bronchitis, pneumonia, pleural effusion or interstitial disease confirmed by chest imaging [X-ray (anteroposterior or anteroposterior) /CT] and judged clinically significant by the investigator at screening.
* 4. Subjects who have developed acute respiratory tract infection, otitis media, and sinusitis within 2 weeks before screening.
* 5. Subjects with other respiratory infections requiring systemic anti-infective treatment, or blood routine examination at screening: white blood cell count (WBC) > (venous blood)
* 6. Subjects with purulent sputum or suppurative tonsillitis.
* 7. Have difficulty in swallowing drugs or have a history of gastrointestinal diseases that seriously affect drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, subtotal gastrectomy, etc.).
* 8. Suspected allergic to active ingredients or excipients of the investigational product.
* 9. Body weight < 20 kg.
* 10. Medications against influenza virus within 7 days before screening (including but not limited to: neuraminidase inhibitors, hemagglutinin inhibitors, M2 ion channel blockers, and cap structure inhibitors. Lysine endonuclease (CEN) inhibitors, such as oseltamivir, zanamivir, peramivir, favipiravir, rimantadine, amantadine, abidol, baloxavir, etc.).
* 11. Have received live vaccines or attenuated live vaccines within 14 days before randomization, influenza vaccines within 6 months before randomization.
* 12. Suspected or confirmed a history of alcohol or drug abuse.
* 13. Ppregnancy test was positive
* 14. Participants who participated in another clinical trial and used any other investigational drug or device within 30 days before screening.
* 15. Subjects judged by the investigator to be ineligible for participation in the study.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of ZX-7101A and its metabolite ZX-7101 in plasma | Part 1: 1~2, 4, 8, 24, 96 ,192, 336 hours post-dose
  Part 1:
  Time to peak drug concentration (Tmax)
Pharmacokinetic parameters of ZX-7101A and its metabolite ZX-7101 in plasma | Part 1: 1~2, 4, 8, 24, 96 ,192, 336 hours post-dose
  Part 1:
  Peak plasma concentration (Cmax)
Pharmacokinetic parameters of ZX-7101A and its metabolite ZX-7101 in plasma | Part 1: 1~2, 4, 8, 24, 96 ,192, 336 hours post-dose
  Part 1:
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic parameters of ZX-7101A and its metabolite ZX-7101 in plasma | Part 1: 1~2, 4, 8, 24, 96 ,192, 336 hours post-dose
  Part 1:
  The terminal elimination half-life (t1/2)
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Part 2: From day1 up to day15
  Part 2:
  The Number of Participants with Treatment-Related Adverse Event will be evalated as the change of vital signs, electrocardiogram, physical examination, and Laboratory test compared with the baseline.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Part 1: From day1 up to day15
  Part 1:
  The Number of Participants with Treatment-Related Adverse Event will be evalated as the change of vital signs, electrocardiogram, physical examination, and Laboratory test compared with the baseline.
Time (in hours) for relief of 7 all influenza symptoms | Part 2: Baseline, Day 1 up to Day 15
  Part 2:
  Symptom remission is defined as a score of 0 (asymptomatic) or 1 (mild) for all seven influenza symptoms assessed by the subject on the subject diary card. And lasts for at least 21.5 hours (approximately 24 hours-10%)
Proportion of all subjects with remission of influenza symptoms | Part 2: Baseline, Day 1 up to Day 15
  Part 2: Proportion of subjects with remission of all influenza symptoms at each visit and each evaluation time point (unit: %);
Influenza virus RNA clearance time (in hours) | Part 2: Baseline, Day1, Day2, Day3, Day5, Day9, Day15
  Part 2: The time to influenza RNA clearance in hours was defined as the time from the start of study treatment to the first time influenza RNA was below the lower limit of quantification (as measured by RT-PCR).
Time for influenza virus titer to become negative | Part 2: Baseline, Day1, Day2, Day3, Day5, Day9, Day15
  Part 2: Time for influenza virus titer to become negative (in hours)
Changes in influenza RNA and virus titers | Part 2: Baseline, Day1, Day2, Day3, Day5, Day9, Day15
  Changes from baseline in RT-PCR-determined influenza RNA (log10 viral copies per milliliter) and virus titers (log10TCID50 per milliliter) at each visit.
Influenza virus RNA | Part 2: Baseline, Day1, Day2, Day3, Day5, Day9, Day15
  Proportion of subjects positive for influenza virus RNA by RT-PCR and with detectable virus titers at each visit (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Liu, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (3):
- China (3):
  - Baoding Hospital of Beijing Children's Hospital, Capital Medical University, Baoding, Hebei
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The results of the trial will be used for New Drug Application.